CLINICAL TRIAL: NCT05462860
Title: Suprathel® Use During Prolonged Field Care to Promote Healing and Reduce the Need for Grafting of Burn Wounds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Metis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Suprathel; CDMRP-MB200024 (Other Grant/Funding Number: Congressionally Directed Medical Research Program Office)
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Wound of Skin; Burns
MeSH Terms: conditions — Burns | interventions — poly(lactide-co-trimethylenecarbonate-co-epsilon-caprolactone); Standard of Care

STUDY DESIGN:
Intervention Model Description: Proof of concept
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suprathel® dressing (Experimental): The Suprathel® dressing will be applied to the wound site after standard of care cleaning and debridement. The dressing will be maintained according to the manufacturer's instructions for use
  Interventions: Other: Suprathel®
- Standard of Care (Active Comparator): The Standard of care as prescribed will be followed for the dressing application for the wound site. Dressings will be applied to the wound site after standard of care cleaning and debridement.
  Interventions: Other: Suprathel®

INTERVENTIONS:
Other: Suprathel® — Application of standard of care dressing.®
  Other Names: standard of care

SUMMARY:
The purpose of this study is to determine the effect to which Suprathel® (Polymedics Innovations GmbH, Denkendorf, Germany) can reduce the need for grafting compared to Standard of Care (SoC). Furthermore, the study intends to evaluate if Suprathel® allows for a reduction of reduction of pain, infection, provider workload, scar development and costs compared to SoC.

DETAILED DESCRIPTION:
We are advocating the study of Suprathel® (Polymedics Innovations GmbH, Denkendorf, Germany), a synthetic wound dressing made of polymers of D-,L- lactate, and ε caprolactone, in the early coverage of burns for use in Large Scale Combat Operations (LSCOs) as compared to standard of care. The rationale for studying Suprathel® is its favorable physical characteristics as a portable treatment, ease of application by personnel without formal medical training, proven efficacy in improving outcomes after partial-thickness burn injury to include better pain control, preliminary evidence in decreasing burn wound conversion, and the lack of adverse consequences in covering indeterminant depth or full thickness burns.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ≥18 years and ≤75 years
* Acute partial thickness burns by friction, contact, scalding from hot liquids and flame
* TBSA total ≥2 %; burn treatment region of interest: all areas with partial-thickness burns excluding face, neck, scalp, and feet
* TBSA 3rd ≤5 % (not to be included as burn treatment region of interest)
* Subject is able and willing to sign Informed Consent or via legally authorized representative

Exclusion Criteria:

* Study Wound due to electrical, radioactive, or frostbite-related injury
* Infection of wounds in the study area at admission per Investigator or treating physician discretion
* Pregnancy/lactation
* Subjects who are unable to follow the protocol or who are likely to be non-compliant
* Participation in an active treatment arm of a burn wound related interventional study within 90 days of Screening Visit or during the study
* Prisoners
* Life expectancy less than 6 months
* Subjects who are receiving steroids, chronic anticoagulants, or immune suppressive treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2025-12-29 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
Need for autograft application | 21 days
  The reduction of need for grafting measured by the percentage of subjects who are converting to grafting at 21 ± 3 days after application.

SECONDARY OUTCOMES:
Wound infection rate, wound closure of the region | 2 weeks, 3 weeks, and 6 weeks after application (without drainage or dressing requirements confirmed at two consecutive study visits 2 weeks apart)
  Incidence of infections and inflammatory response and scar development
Mid and long term clinical scar maturation assessed by the Patient and Observer Scar Assessment Scale (POSAS). | Mid (3-9 months) and long term (52 weeks)
  Patient and Observer Scar Assessment Scale (POSAS) Questionnaire is used to assess scarring.
Patient-reported perception of pain based on the Visual Analog Scale | After initial application (Day 0) and weekly
  Patients will be asked to rate their pain 0-10 (0=no pain and 10=a lot of pain) prior to and after application of the first dressing and subsequent dressings.

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Chan, MD, Principal Investigator — Metis Foundation
Locations (1):
- North Carolina Jaycee Burn Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No